CLINICAL TRIAL: NCT03813251
Title: Safety and Effectiveness Evaluation of the ForConti Contix Fecal Incontinence Management System (FIMS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ForConti Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-14-002
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Assigned Interventions (Experimental): ForConti Contix Fecal Incontinence Management System (FIMS)
  Interventions: Device: ForConti Contix Fecal Incontinence Management System (FIMS)

INTERVENTIONS:
Device: ForConti Contix Fecal Incontinence Management System (FIMS) — Use the device for up to 12 hours per use for 4 weeks

SUMMARY:
The ForConti Contix Fecal Incontinence Management System (FIMS) is indicated for the management of accidental bowel leakage due to bowel incontinence. The ForConti Contix FIMS is designed to seal and help prevent the involuntary leakage of stool, liquids and gases from the rectum. ForConti Contix FIMS is for an individual with fecal incontinence that has impaired quality of life, is responsive and mentally capable to participate in their own treatment.

This study is designed to evaluate the safety and effectiveness of the ForConti Contix FIMS for its intended use utilizing a baseline period of 2 weeks followed by an on-device period of using the device for 4 weeks and completed with a followup period of 2 weeks.

DETAILED DESCRIPTION:
Treatments for bowel incontinence depend on the cause and severity of the condition. Often more than one modality is used to treat the condition, beginning with conservative options such as adult diapers and pads, medication, biofeedback and anal plugs/balloons and moving on to invasive procedures (i.e. nerve stimulators, restorative surgery, colostomy) where conservative treatment isn't effective.

The main reason for potential pain and discomfort with the current available anal plugs is the plug location within the anus below the dentate line. This part of the anus, which is highly sensitive, may cause discomfort and pain to some users. The advantage of the ForConti Contix Fecal Incontinence Management System (FIMS) is that it is designed to be located in an inner section of the rectum, above the dentate line, and therefore less sensitive and less likely to cause discomfort or pain to the user.

This study is a prospective, non-randomized, single-arm, self-controlled clinical investigation designed to evaluate the safety and effectiveness of the ForConti Contix FIMS. Total duration of the study for each patient will be 8 weeks, including follow-up.

This multi center study will be conducted on 10-20 patients (per site) suffering from accidental bowel leakage due to bowel incontinence and who meet all of the inclusion criteria and none of the exclusion criteria.

The ForConti Contix FIMS includes 2 main parts: the inserted part and the insertion system. The inserted part includes a balloon and a pulling string, and the insertion system includes the applicator and the inflation kit. The balloon is a soft flexible biocompatible, component. It is designed to be located in the rectum by an applicator and to be filled with a pre-determined amount of air to gain its final shape.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the informed consent form and is willing to participate in the clinical study. Patient has the ability to self-manage insertion and removal of the device
2. Patient age is between 22 and 85 years old
3. Patient has history of fecal incontinence for at least 6 months
4. Patient has a minimum of four incontinence episodes during the 2-week baseline period
5. Patient colon surveillance complies with National Program/Guidelines for the Early Detection of Colorectal Cancer
6. Patient comprehends study meaning and is capable of carrying out study duties
7. If the candidate is currently prescribed medication per os or per rectum for bowel control, treatment has been administered for at least 4 weeks without a change in treatment regimen or dose, and the candidate agrees to continue the treatment without changes for the duration of the study

Exclusion Criteria:

1. Patient had spinal cord injury or other major neurological diagnosis
2. Patient has known life threatening disease such as cancer, immune deficiency state
3. Patient has significant cardiac arrhythmia*
4. Patient has inflammatory bowel disease
5. Patient is on anti-coagulants and anti-platelets treatment, except Aspirin (low dose: 75-100 mg/day)
6. Patient has anorectal disease: perianal abscess, active fistula, fissure, hemorrhoids grade 3 or 4, Pruritus ani or rectal bleeding*
7. Patient has a clinically significant abnormality as visualized by sigmoidoscopy at the first visit
8. Patient has pre-existing rectal pain or rectal bleeding
9. Patient suffers from chronic pelvic pain
10. Patient had rectal surgery in the past 6 months
11. Patient has rectocele or other pelvic organ prolapse requiring surgery*
12. Patient has allergy to silicone or one of its components
13. Patient has significant medical condition which may interfere with study participation
14. Patient is currently participating in another clinical study.
15. Female patient is pregnant or breastfeeding

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Number of device related serious adverse events | 6 weeks (4 weeks of use and 2 weeks follow-up)
  Number of device related serious adverse events
Rate of subjects who improved by 50% or more in ABL (FI episodes) during the on-device period as compared to the baseline period. | 8 weeks (2 weeks baseline, 4 weeks of use and 2 weeks follow-up)
  ≥40% of subjects reporting ≥50% reduction in FI episodes during the on-device period as compared to the baseline period.

SECONDARY OUTCOMES:
Rate of device or procedure related adverse events in the treatment or in the follow-up periods. | 6 weeks (4 weeks of use and 2 weeks follow-up)
  Rate of device or procedure related adverse events in the treatment or in the follow-up periods.
Change in mean scores on subject-reported outcomes related to symptom-specific Fecal Incontinence Quality of Life (FIQoL) Questionnaire. | 6 weeks (2 weeks baseline, 4 weeks of use )
  Fecal Incontinence Quality of Life scale (all subscale scores 1-4) Scales range from 1 to 5, with a 1 indicating a lower functional status of quality of life. Scale scores are the average (mean) response to all items in the scale (e.g., add the responses to all questions in a scale together and then divide by the number of items in the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy B Menees, MD, Principal Investigator — University of Michigan, Department of Medicine, Division of Gastroenterology; William D Chey, MD, Principal Investigator — University of Michigan, GI Physiology Laboratory; Lin Chang, MD, Principal Investigator — David Gefen School of Medicine at UCLA, Division of Digestive Diseases

IPD SHARING:
Plan to Share IPD: No